CLINICAL TRIAL: NCT01183689
Title: Study of Novel Approaches for Prevention
Acronym: SNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00010097; 5U01HL090875 (NIH)
Record Dates: First submitted 2010-08-13; First posted 2010-08-18 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): "Self-Guided Behavior Changes". This group will be used to determine average rate of weight gain over 3 years with little intervention. Participants randomized to this group will receive one face-to-face session that will provide general education of self-weighing and information about both the small and large changes approach. Participants will also be provided with quarterly newsletters describing study events and very limited information on health eating.
- Small behavior changes (Experimental): Participants randomized to this group will be taught to self-weigh daily and report weights regularly. They will be reinforced for maintaining weight below randomization weight and taught that if weight exceeds randomization weight, they should reinstate small changes (e.g., modify diet by approximately 100 kcal, decrease portion sizes or change types of food, increase activity by 2000 steps/day).
  Interventions: Behavioral: Small Behavior Changes
- Large behavior changes (Experimental): Participants randomized to this group will be taught to self-weigh daily and report weights regularly. They will be reinforced for maintaining weight below randomization weight and taught that if weight exceeds randomization weight, they should reinstate large changes (e.g., modify diet to 1200-1500 or 1500-1800 kcal/day with < 30% fat, increase exercise to 250 minutes/week of moderate intensity activity).
  Interventions: Behavioral: Large Behavior Changes

INTERVENTIONS:
Behavioral: Small Behavior Changes — The Self-Regulation Plus Small Behavior Changes Intervention will focus on making small changes in diet and physical activity on a daily basis to prevent weight gain.
  Diet: The dietary approach used in this group is to identify small changes in what and how much participants eat each day. The general concept is that these are small, manageable changes that will produce small reductions in overall intake and can easily be made on a daily basis and maintained over time.
  Exercise: At the start of the program, participants will be given a pedometer and asked to record their current or baseline number of steps. They will then be given the goal of increasing their daily steps by 2000 steps per day over this baseline level.
  Other Names: Small Behavior Changes plus self-regulation
  Arms: Small behavior changes
Behavioral: Large Behavior Changes — The focus of this intervention group will be on periodically making large changes in diet and physical activity, with the goal of losing 5-10 pounds to buffer against the weight gain that often occurs during young adulthood.
  Diet: Individuals with a BMI of 21-24.9 kg/m2 will be encouraged to lose 5 pounds; those with a BMI of 25-30 kg/m2 will be encouraged to lose 10 pounds.
  Exercise: The Large Changes group will be instructed to gradually increase their minutes of physical activity until achieving 250 minutes per week (5 days/week with 50 minutes per day) using activities similar in intensity to brisk walking.
  Other Names: Large Behavior Changes plus self-regulation
  Arms: Large behavior changes

SUMMARY:
The Study of Novel Approaches for Prevention (SNAP) is randomized trial designed to test whether behavioral interventions based on self-regulation can prevent weight gain in young adults (18-35 years; body mass index (BMI) 21-30 kg/m2). Two different self-regulation interventions for weight gain prevention will be compared in this trial; one intervention will focus on making small, consistent, changes in eating and exercise behavior to prevent weight gain or reverse weight gain if it occurs, whereas the other will emphasize larger changes in eating and exercise that occur periodically, with a goal of producing weight loss and thereby providing a buffer against anticipated weight gains. The primary aim of the trial is to test whether the magnitude of weight gain from baseline across an average three-year follow-up differs across the three groups, with the hypotheses that weight gain will be greater in the Control group than in either intervention and greater in the Small Changes than Large Changes group.

SNAP-E (Extension) will determine whether the effects of the intervention can be maintained over an additional 3 years (i.e. through a total of 6 years).

DETAILED DESCRIPTION:
Young adults, aged 20-35 years, experience the greatest rate of weight gain, averaging 1-2 lbs/yr. Over time, this weight gain is associated with a worsening in cardiovascular disease risk factors and an increase in the prevalence of metabolic syndrome. Given the difficulties in producing sustained weight loss later in life, preventing weight gain from occurring during this critical period is key to curbing the obesity epidemic. The Study of Novel Approaches for Prevention (SNAP) is a 2-center randomized trial designed to test whether behavioral interventions based on self-regulation can prevent weight gain in young adults (18-35 years; body mass index (BMI) 21-30 kg/m2). Approximately 600 participants will be recruited over two years and randomly assigned to a control condition (N=200), self-regulation with small changes (N=200) or self-regulation with large changes (N=200). The Small Changes group will be taught to make small, consistent, changes in eating and exercise behavior to prevent weight gain or reverse weight gain if it occurs whereas the Large Changes group will emphasize periodic, larger changes in eating and exercise, with a goal of producing weight loss and thereby providing a buffer against anticipated weight gain. The primary aim of the trial is to test whether the magnitude of weight gain from baseline across an average planned follow-up of three years differs across the three groups, with a priori hypotheses that weight gain will be greater in the Control group than in either intervention and greater in the Small Changes than Large Changes group. Secondary aims are to compare the three groups on a) the proportion of participants in the three groups who gain less than 1 pound over the planned follow-up, b) the mean difference in weight gain from baseline to 24-month follow-up, c) the changes in behaviors and psychosocial measures (diet, physical activity, dietary restraint, frequency of self-weighing,depression, and occurrence of abnormal eating behaviors), and d) the changes in cardiovascular disease risk factors (blood pressure, lipids, insulin sensitivity, and waist circumference). The trial will also examine the association among changes in behaviors, weight, and cardiovascular disease risk factors and examine variables that may moderate the effects of the intervention (including gender, ethnicity, initial BMI, age) and potential mediators of the effects of the intervention (including changes in diet, activity, and self-regulatory behaviors). SNAP is member of the Early Adult Reduction in Weight Through Lifestyle Interventions (EARLY) consortium of clinical trials funded by the National Heart, Lung, and Blood Institute.

ELIGIBILITY:
Inclusion Criteria:

1. BMI of 21 - 30 kg/m2

Exclusion Criteria:

1. Untreated hypertension, hyperlipidemia, or type 2 diabetes, unless permission is provided by their health care provider.
2. Heart disease, heart problems or report being prescribed drugs for blood pressure or a major heart condition, unless permission is provided by their health care provider.
3. Type 1 diabetes or treatment of type 2 diabetes with insulin or oral medication that may cause hypoglycemia.
4. Health problems which may influence the ability to walk for physical activity (e.g. lower limb amputation) or other reasons why a person should not do physical activity, unless permission is provided from their health care provider.
5. Health problems that may be associated with unintentional weight change or affect the safety of a weight loss program, including report of a heart attack or stroke, chest pain during periods of activity or rest, loss of consciousness, active tuberculosis, HIV, chronic hepatitis B or C, inflammatory bowel disease requiring treatment within the past year, thyroid disease, renal disease, liver disease, hospitalization for asthma in the past year, or cancer within the past 5 years (except for non-melanoma skin cancers or early stage cervical cancer) or chronic use of steroid medication.
6. Report of a past diagnosis of or treatment for a Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision (DSM-IV-TR) eating disorder (anorexia nervosa or bulimia nervosa) or meet criteria for anorexia or bulimia nervosa during screening for this trial
7. Report of a past diagnosis of or current symptoms of alcohol or substance dependence.
8. Currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 6 months.
9. History of schizophrenia, manic depression, or bipolar disorder.
10. Hospitalization for depression or other psychiatric disorder within the past 12 months.
11. Having lost and maintained a weight loss of 10 pounds or more within the past 6 months or are currently participating in a weight loss program, trying to gain weight, using steroids for muscle mass or weight gain, taking weight loss medication, or have had surgery for weight loss.
12. Participation in another weight loss or physical activity study that would interfere with this study.
13. Another member of the household (or roommate) is a participant or staff member on this trial.
14. Reason to suspect that the participant would not adhere to the study intervention or assessment schedule (i.e., can't come to group on a regular basis; will be away for more than two weeks during initial intervention phase or planning to move from the area within next year).
15. Not able to speak and understand English.
16. Residence or place of work further than 30 miles from the intervention site.
17. Perceived inability to attend the 2 year data collection visit.
18. Does not have Internet access on a regular basis.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 599 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rena Wing, PhD, Study Chair — The Miriam Hospital; Judy Bahnson, Principal Investigator — Wake Forest University Health Sciences; Wei Lang, PhD, Principal Investigator — Wake Forest University Health Sciences; Mark A Espeland, PhD, Principal Investigator — Wake Forest University Health Sciences; Deborah Tate, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Beth Lewis, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
De-identified data can be obtained by request, conditional on a data use agreement.

REFERENCES:
- [Derived] Hayes JF, LaRose JG, Gorin AA, Lewis CE, Bahnson J, Phelan S, Wing RR; Study of Novel Approaches to Weight Gain Prevention (SNAP) Research Group. Weight gain prevention interventions in the Study of Novel Approaches to Weight Gain Prevention (SNAP) trial promote ideal cardiovascular health in young adults. Obesity (Silver Spring). 2023 Jun;31(6):1530-1537. doi: 10.1002/oby.23753. Epub 2023 May 8. PMID 37157110
- [Derived] Corso LML, Wing RR, Tate DF, Espeland MA, Blanchard BE, McCaffery JM. Uric acid as a predictor of weight gain and cardiometabolic health in the Study of Novel Approaches to Weight Gain Prevention (SNAP) study. Int J Obes (Lond). 2022 Aug;46(8):1556-1559. doi: 10.1038/s41366-022-01131-1. Epub 2022 May 2. PMID 35501471
- [Derived] Wing RR, Espeland MA, Tate DF, Perdue LH, Bahnson J, Polzien K, Robichaud EF, LaRose JG, Gorin AA, Lewis CE, Jelalian E; Study of Novel Approaches to Weight Gain Prevention (SNAP) Research Group. Weight Gain Over 6 Years in Young Adults: The Study of Novel Approaches to Weight Gain Prevention Randomized Trial. Obesity (Silver Spring). 2020 Jan;28(1):80-88. doi: 10.1002/oby.22661. PMID 31858732
- [Derived] LaRose JG, Neiberg RH, Evans EW, Tate DF, Espeland MA, Gorin AA, Perdue L, Hatley K, Lewis CE, Robichaud E, Wing RR; Study of Novel Approaches to Weight Gain Prevention (SNAP) Research Group. Dietary outcomes within the study of novel approaches to weight gain prevention (SNAP) randomized controlled trial. Int J Behav Nutr Phys Act. 2019 Jan 31;16(1):14. doi: 10.1186/s12966-019-0771-z. PMID 30704533
- [Derived] Olson KL, Neiberg RH, Tate DF, Garcia KR, Gorin AA, Lewis CE, Unick J, Wing RR. Weight and Shape Concern Impacts Weight Gain Prevention in the SNAP Trial: Implications for Tailoring Intervention Delivery. Obesity (Silver Spring). 2018 Aug;26(8):1270-1276. doi: 10.1002/oby.22212. Epub 2018 Jun 28. PMID 29956495
- [Derived] McCaffery JM, Ordovas JM, Huggins GS, Lai CQ, Espeland MA, Tate DF, Wing RR. Weight gain prevention buffers the impact of CETP rs3764261 on high density lipoprotein cholesterol in young adulthood: The Study of Novel Approaches to Weight Gain Prevention (SNAP). Nutr Metab Cardiovasc Dis. 2018 Aug;28(8):816-821. doi: 10.1016/j.numecd.2018.02.018. Epub 2018 Mar 6. PMID 29699816
- [Derived] Unick JL, Lang W, Williams SE, Bond DS, Egan CM, Espeland MA, Wing RR, Tate DF; SNAP Research Group. Objectively-assessed physical activity and weight change in young adults: a randomized controlled trial. Int J Behav Nutr Phys Act. 2017 Dec 4;14(1):165. doi: 10.1186/s12966-017-0620-x. PMID 29202850
- [Derived] Wing RR, Tate DF, Garcia KR, Bahnson J, Lewis CE, Espeland MA; Study of Novel Approaches to Weight Gain Prevention (SNAP) Research Group. Improvements in Cardiovascular Risk Factors in Young Adults in a Randomized Trial of Approaches to Weight Gain Prevention. Obesity (Silver Spring). 2017 Oct;25(10):1660-1666. doi: 10.1002/oby.21917. Epub 2017 Aug 7. PMID 28782918
- [Derived] Unick JL, Lang W, Tate DF, Bond DS, Espeland MA, Wing RR. Objective Estimates of Physical Activity and Sedentary Time among Young Adults. J Obes. 2017;2017:9257564. doi: 10.1155/2017/9257564. Epub 2017 Jan 2. PMID 28116151
- [Derived] Crane MM, LaRose JG, Espeland MA, Wing RR, Tate DF. Recruitment of young adults for weight gain prevention: randomized comparison of direct mail strategies. Trials. 2016 Jun 8;17(1):282. doi: 10.1186/s13063-016-1411-4. PMID 27278474
- [Derived] Wing RR, Tate DF, Espeland MA, Lewis CE, LaRose JG, Gorin AA, Bahnson J, Perdue LH, Hatley KE, Ferguson E, Garcia KR, Lang W; Study of Novel Approaches to Weight Gain Prevention (SNAP) Research Group. Innovative Self-Regulation Strategies to Reduce Weight Gain in Young Adults: The Study of Novel Approaches to Weight Gain Prevention (SNAP) Randomized Clinical Trial. JAMA Intern Med. 2016 Jun 1;176(6):755-62. doi: 10.1001/jamainternmed.2016.1236. PMID 27136493
- [Derived] Wing RR, Tate D, LaRose JG, Gorin AA, Erickson K, Robichaud EF, Perdue L, Bahnson J, Espeland MA. Frequent self-weighing as part of a constellation of healthy weight control practices in young adults. Obesity (Silver Spring). 2015 May;23(5):943-9. doi: 10.1002/oby.21064. Epub 2015 Apr 10. PMID 25865175
- [Derived] Tate DF, LaRose JG, Griffin LP, Erickson KE, Robichaud EF, Perdue L, Espeland MA, Wing RR. Recruitment of young adults into a randomized controlled trial of weight gain prevention: message development, methods, and cost. Trials. 2014 Aug 16;15:326. doi: 10.1186/1745-6215-15-326. PMID 25128185
- [Derived] Wing RR, Tate D, Espeland M, Gorin A, LaRose JG, Robichaud EF, Erickson K, Perdue L, Bahnson J, Lewis CE. Weight gain prevention in young adults: design of the study of novel approaches to weight gain prevention (SNAP) randomized controlled trial. BMC Public Health. 2013 Apr 4;13:300. doi: 10.1186/1471-2458-13-300. PMID 23556505

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SNAP targeted an enrollment of 600 participants, aged 18-35 years, with a BMI of 21.0 to 30.9. Participants were recruited from 2 clinical sites (Providence, RI and Chapel Hill, NC). The final sample of 599 participants (27% minority, 22% male) was recruited over a 19-month period (Aug 2010-Feb 2012).
Pre-assignment Details: Participants were pre-screened online and by telephone before attending an orientation, followed by two screening visits. 609 participants were randomized; although 10 participants never attended the randomization visit and did not learn of their group assignment.
Groups:
- Self-regulation With Small Behavior Changes: Participants randomized to this group will be taught to self-weigh daily and report weights regularly. They will be reinforced for maintaining weight below randomization weight and taught that if weight exceeds randomization weight, they should reinstate small changes (e.g., modify diet by approximately 100 kcal, decrease portion sizes or change types of food, increase activity by 2000 steps/day).
  Self-regulation theory: Participants randomized to either of these two groups will be taught to self-weigh daily and report weights regularly. They will be reinforced for maintaining weight below randomization weight and taught that if weight exceeds randomization weight, they should reinstate either large or small changes.
- Self-regulation With Large Behavior Changes: Participants randomized to this group will be taught to self-weigh daily and report weights regularly. They will be reinforced for maintaining weight below randomization weight and taught that if weight exceeds randomization weight, they should reinstate large changes (e.g., modify diet to 1200-1500 or 1500-1800 kcal/day with < 30% fat, increase exercise to 250 minutes/week of moderate intensity activity).
  Self-regulation theory: Participants randomized to either of these two groups will be taught to self-weigh daily and report weights regularly. They will be reinforced for maintaining weight below randomization weight and taught that if weight exceeds randomization weight, they should reinstate either large or small changes.
Period: Overall Study
Arm/Group | Control Group | Self-regulation With Small Behavior Changes | Self-regulation With Large Behavior Changes
Started | 202 | 200 | 197
Month 4 Visit | 197 | 192 | 187
Year 1 Visit | 187 | 172 | 183
Year 2 Visit | 178 | 172 | 174
Year 3 Visit | 139 | 125 | 126
Year 4 Visit | 38 | 33 | 30
Completed | 202 | 200 | 197
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Self-regulation With Small Behavior Changes | Self-regulation With Large Behavior Changes | Total
Number analyzed (Participants) | 202 | 200 | 197 | 599
Age, Customized [Count of Participants; unit: Participants]
  Age: Age : 18-24 years | 53 | 60 | 56 | 169
  Age: Age : 25-35 years | 149 | 140 | 141 | 430
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 157 | 154 | 469
  Male | 44 | 43 | 43 | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American | 19 | 25 | 22 | 66
  Race/Ethnicity: Non-Hispanic white | 148 | 146 | 144 | 438
  Race/Ethnicity: Asian/Pacific Islander | 7 | 11 | 7 | 25
  Race/Ethnicity: Hispanic | 15 | 10 | 21 | 46
  Race/Ethnicity: Multiple/Refused | 13 | 8 | 3 | 24
BMI [Count of Participants; unit: Participants]
  <25.0 kg/m2 | 97 | 84 | 96 | 277
  >=25.0 kg/m2 | 105 | 116 | 101 | 322
Weight [Mean (Standard Deviation); unit: kilograms] | 71.4 (10.2) | 71.9 (11.0) | 70.8 (11.0) | 71.4 (10.7)
Education [Count of Participants; unit: Participants]
  Not college graduate | 39 | 46 | 35 | 120
  College graduate | 163 | 154 | 162 | 479
Employment Status [Count of Participants; unit: Participants]
  Employed full time | 127 | 125 | 125 | 377
  Student full time | 49 | 61 | 55 | 165
  Other | 26 | 14 | 17 | 57

OUTCOME MEASURES:

1. Primary Outcome: Weight Changes From Baseline Over Follow-up.
Description: Mean weight change from baseline across an average planned follow-up of three years. These mean changes will be compared among the three arms of the trial.
Time Frame: 3 years
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Control Group | Self-regulation With Small Behavior Changes | Self-regulation With Large Behavior Changes
Number analyzed (Participants) | 202 | 200 | 197
kilograms | 0.26 (0.22) | -0.56 (0.22) | -2.37 (0.22)
Statistical Analysis 1: Comparison: Control Group vs Self-regulation With Small Behavior Changes; Mean changes from random effects model applied to repeated measures to compute the average differences among groups over time; Test type: Superiority; p < 0.05, Mixed Models Analysis — No interim analyses were conducted. Pairwise differences among the three arms were assessed with a 2 degree of freedom Wald Test; Mean Difference (Net) = 0.82, 95% CI 2-sided [0.23 to 1.41], Standard Error of Mean 0.30 — Above is provided the mean difference between Arms 1 and 2
Statistical Analysis 2: Comparison: Control Group vs Self-regulation With Large Behavior Changes; Mean changes from a random effects model applied to repeated measures to compute the average differences between groups over time. This entry is for the comparison between groups 1 and 3; Test type: Superiority; p < 0.05, Mixed Models Analysis; This was fitted with Proc Mixed in SAS; Mean Difference (Net) = 2.64, 95% CI 2-sided [2.05 to 3.22] — 95% confidence interval excludes 0

2. Secondary Outcome: Weight Gain 1 Pound or More at Any Time Over Follow-up
Description: Average over time (average follow-up of 3 years) of the percent of participants within each arm of the trial who gain 1 pound or more at each visit. These percentages will be compared among the three arms generalized estimating equations. Note that weight changes in units of pounds were used to define this outcome so that it may be more clear to participants. Elsewhere in the protocol, weight is reported in kilograms. Percentages at each visit are the percent who gained 1 pound or more from baseline among all who were weighed at that visit. Participants were assigned values of 0 or 1 at each visit depending on their weight gain status.
Time Frame: 3 years
Measure: Mean (Standard Error); unit: percentage gaining 1 pound or more among
Arm/Group | Control Group | Self-regulation With Small Behavior Changes | Self-regulation With Large Behavior Changes
Number analyzed (Participants) | 202 | 200 | 197
percentage gaining 1 pound or more among | 40.8 (4.4) | 32.5 (3.8) | 23.6 (2.8)
Statistical Analysis 1: Comparison: Control Group vs Self-regulation With Small Behavior Changes; Generalized estimating equations were used to compare the average percent of weight gainers over time among the three groups. The null hypothesis was that there was no difference in these average percentages. Participants were assigned values of 0 or 1 at each visit depending on their weight gain status. The percentages were summarized with odds ratios for weight gain over time; Test type: Other — Generalized Estimating Equations; p < 0.05, Generalized Estimating Equations; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.02 to 1.90]
Statistical Analysis 2: Comparison: Control Group vs Self-regulation With Large Behavior Changes; This is a parallel analysis, comparing groups 1 and 3, using generalized estimating equations to summarize the odds ratio for weight gain in group 1 versus group 3,; Test type: Superiority; p < 0.05, generalized estimating equations; Odds Ratio (OR) = 2.28, 95% CI 2-sided [1.64 to 3.19]

3. Secondary Outcome: Mean Weight Changes
Description: Mean differences in weight changes among intervention groups at 24 months post-randomization
Time Frame: 2 years
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Control Group | Self-regulation With Small Behavior Changes | Self-regulation With Large Behavior Changes
Number analyzed (Participants) | 202 | 200 | 197
kilograms | 0.54 (0.33) | -0.77 (0.33) | -1.50 (0.34)
Statistical Analysis 1: Comparison: Control Group vs Self-regulation With Small Behavior Changes; Mean differences at 2 years are calculated from a linear contrast within a mixed effects model. Note that this comparison is between Groups 1 and 2; Test type: Superiority; p < 0.05, Mixed Models Analysis; The p-value is based on a 2 degree of freedom Wald test within the mixed effect model to test for pairwise differences among the 3 arms; Mean Difference (Net) = 1.31, 95% CI 2-sided [0.39 to 2.24], Standard Error of Mean 0.47 — Listed above is the mean difference between arms 1 and 2
Statistical Analysis 2: Comparison: Control Group vs Self-regulation With Large Behavior Changes; A linear contrast from a mixed effects model was used to compare mean differences at 24 months between groups 1 and 3; Test type: Superiority; p < 0.05, Mixed Models Analysis; A linear contrast was used to compare groups 1 and 3 at 24 months; Median Difference (Net) = 2.04, 95% CI 2-sided [1.11 to 2.98]

4. Secondary Outcome: Mean Changes in Systolic Blood Pressure
Description: Compare changes in systolic blood pressure across the three intervention groups
Time Frame: Measured at 2 Years
Population: All participants with measurements at Year 2
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Small Behavior Changes: Participants randomized to this group will be taught to self-weigh daily and report weights regularly. They will be reinforced for maintaining weight below randomization weight and taught that if weight exceeds randomization weight, they should reinstate small changes (e.g., modify diet by approximately 100 kcal, decrease portion sizes or change types of food, increase activity by 2000 steps/day).
  Small Behavior Changes: The Self-Regulation Plus Small Behavior Changes Intervention will focus on making small changes in diet and physical activity on a daily basis to prevent weight gain.
  Diet: The dietary approach used in this group is to identify small changes in what and how much participants eat each day. The general concept is that these are small, manageable changes that will produce small reductions in overall intake and can easily be made on a daily basis and maintained over time.
  Exercise: At the start of the program, participants will be given a pedometer and asked
- Large Behavior Changes: Participants randomized to this group will be taught to self-weigh daily and report weights regularly. They will be reinforced for maintaining weight below randomization weight and taught that if weight exceeds randomization weight, they should reinstate large changes (e.g., modify diet to 1200-1500 or 1500-1800 kcal/day with < 30% fat, increase exercise to 250 minutes/week of moderate intensity activity).
  Large Behavior Changes: The focus of this intervention group will be on periodically making large changes in diet and physical activity, with the goal of losing 5-10 pounds to buffer against the weight gain that often occurs during young adulthood.
  Diet: Individuals with a BMI of 21-24.9 kg/m2 will be encouraged to lose 5 pounds; those with a BMI of 25-30 kg/m2 will be encouraged to lose 10 pounds.
  Exercise: The Large Changes group will be instructed to gradually increase their minutes of physical activity until achieving 250 minutes per week (5 days/week with 50 minutes
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 158 | 154 | 159
mmHg | 1.73 (0.69) | -3.72 (0.70) | -2.66 (0.69)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Analysis of variance to assess mean differences in changes from baseline in systolic blood pressure. This analysis compares groups 1 and 2; Test type: Superiority; p = 0.13, ANOVA — The p-value is from a 2 degree of freedom test for pairwise difference among the 3 arms within an analysis of variance; Mean Difference (Net) = 1.99, 95% CI 2-sided [0.06 to 3.92]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Mean differences in systolic blood pressure between groups 1 and 3 over time; Test type: Superiority; p = 0.13, ANOVA; Mean Difference (Net) = 0.93, 95% CI 2-sided [-0.98 to 2.84]

5. Secondary Outcome: Mean Changes From Baseline in Diastolic Blood Pressure
Description: Change from baseline to 2 years in diastolic blood pressure
Time Frame: 2 years
Population: All participants providing data at 2 years
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 158 | 154 | 159
mmHg | -0.41 (0.51) | -2.14 (0.52) | -1.33 (0.51)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Mean differences from baseline to 2 years were compared among the 3 arms using analysis of variance; Test type: Superiority; p = 0.06, ANOVA — The p-value is from a 2 degree of freedom F-test from an analysis of variance to compare mean differences among the 3 arms; Mean Difference (Net) = 1.73, 95% CI 2-sided [0.32 to 3.14]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare mean changes from baseline to 2 years in diastolic blood pressure; Test type: Superiority; p = 0.06, ANOVA — This p-value is from a 2 degree of freedom omnibus test for differences among the 3 groups; Mean Difference (Net) = 0.92, 95% CI 2-sided [-0.49 to 2.33]

6. Secondary Outcome: Mean Changes From Baseline to 2 Years in Total Cholesterol
Description: Mean changes from baseline to 2 years in total cholesterol among participants with Year 2 measurements (mg/dl)
Time Frame: 2 years
Population: All participants with Year 2 measures
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 158 | 154 | 159
mg/dl | -0.56 (1.75) | 0.74 (1.73) | 1.33 (1.75)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Mean changes from baseline to 2 years were compared between Groups 1 and 2; Test type: Superiority; p = 0.73, ANOVA — The p-value results from a 2 degree of freedom F-test; Mean Difference (Net) = -1.30, 95% CI 2-sided [-6.12 to 3.52]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare mean differences in total cholesterol changes from baseline among groups; Test type: Superiority; p = 0.73, ANOVA — This p-value is from a 2 degree of freedom test for differences among the 3 groups; Mean Difference (Net) = -1.89, 95% CI 2-sided [-4.36 to 0.58]

7. Secondary Outcome: Obesity
Description: Percentage of those participants whose body mass index at baseline was less than 30 kg/m2 who subsequently transitioned to a body mass index of 30 kg/m2 or more (i.e. met criteria for obesity) sometime during 3 years of follow-up (i.e. at least one visit). Percentages will be compared among the three arms of the trial and summarized with odds ratios Participants were assigned values of 0 or 1 at each exam depending on their obesity level. Inference is based on generalized estimating equations.
Time Frame: 3 years
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | Control Group | Self-regulation With Small Behavior Changes | Self-regulation With Large Behavior Changes
Number analyzed (Participants) | 195 | 195 | 193
percentage of participants | 16.9 (2.7) | 7.9 (2.0) | 8.6 (2.0)
Statistical Analysis 1: Comparison: Control Group vs Self-regulation With Small Behavior Changes; The average percentage of participants who were obese across follow-up were compared among the 3 arms using a generalized estimating equations approach for repeated binary measures. Participants were assigned values of 0 or 1 depending on their obesity status at each exam. Differences were summarized with odds ratios; Test type: Superiority; p < 0.001, generalized estimating equations — The p-value is a 2 degree of freedom test from the generalized estimating equations analysis applied to the longitudinal binary data among the 3 study arms; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.23 to 4.52]
Statistical Analysis 2: Comparison: Control Group vs Self-regulation With Large Behavior Changes; Generalized estimating equations were used. Differences were summarized with odds ratios; Test type: Superiority; p = 0.008, generalized estimating equations — This p-value is from a 2 degree of freedom test for differences among the 3 groups; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.12 to 4.10]

8. Secondary Outcome: Dietary Restraint: Mean Change From Baseline to 2 Years
Description: The Eating Inventory (Stunkard, 1988) is a 51-item self-report instrument, was used to assess the subscale of dietary restraint (e.g., degree of conscious control exerted over eating behaviors; range from 0-21 with higher scores reflecting greater levels of restraint).
  Reference: Stunkard, A. J. M., S. (1988). Eating Inventory Manual. New York: Psychological Corporation.
Time Frame: 2 years
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 178 | 172 | 174
Units on a scale | 0.39 (0.18) | 0.59 (0.19) | 1.27 (0.19)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Mean changes from baseline to 2 years among the 3 groups were assessed using a 2 degree of freedom F-test; Test type: Superiority; p = 0.002, ANOVA — the p-value results from a 2 degree of freedom F-test to assess pairwise differences among the 3 groups; the p-value results from a 2 degree of freedom F-test to assess pairwise differences among the 3 groups; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.61 to 0.45]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Differences among the 3 groups were based on analyses of variance; Test type: Superiority; p = 0.002, ANOVA — This p-value is from a 2 degree of freedom test for differences among all 3 groups; Mean Difference (Net) = 0.55, 95% CI 2-sided [0.02 to 1.08]

9. Secondary Outcome: Disinhibition
Description: The Eating Inventory (TFEQ(Stunkard, 1988), a 51-item self-report instrument, was used to assess the subscale of disinhibition (e.g., susceptibility to loss of control over eating; range 0-16, with higher scores reflecting greater levels of disinhibition).
  REF: Stunkard, A. J. M., S. (1988). Eating Inventory Manual. New York: Psychological Corporation.
Time Frame: Changes at 2 years
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 178 | 172 | 174
Units on a scale | 0.07 (0.17) | -0.78 (0.17) | -0.03 (0.17)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Changes in units of the scale from baseline to 2 years; Test type: Superiority — A 2 degree of freedom F-test from ANOVA was used to compare mean differences in changes among the 3 arms of the study; p < 0.001, ANOVA — The p-value is from a 2 degree of freedom F test to assess differences among the 3 arms of the study; The p-value is from a 2 degree of freedom F test to assess differences among the 3 arms of the study; Mean Difference (Net) = -0.85, 95% CI 2-sided [-1.32 to -0.38]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare mean changes from baseline to 2 years among the 3 groups; Test type: Superiority; p < 0.001, ANOVA — This p-value is from a 2 degree of freedom test to compare differences among the 3 groups; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.57 to 0.37]

10. Secondary Outcome: Flexible Dietary Control
Description: Flexible control is characterized by a balanced approach to eating (e.g., taking smaller portions to control weight, engaging in healthy compensation) and is associated with better weight management outcomes (Westenhoefer, Stunkard, & Pudel, 1999). Scores range from 0 to 12 with higher scores reflecting greater levels of flexible control.
  REF: Westenhoefer, J., Stunkard, A. J., & Pudel, V. (1999). Validation of the flexible and rigid control dimensions of dietary restraint. Int J Eat Disord, 26(1), 53-64.
Time Frame: Changes from baseline to 2 years
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 178 | 172 | 174
units on a scale | 0.39 (0.18) | 0.59 (0.19) | 1.27 (0.19)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes vs Large Behavior Changes; 2 degree of freedom F-test from analysis of variance to compare 2 year differences from baseline among the 3 arms of the study; Test type: Superiority — 2 degree of freedom F-test from analysis of variance to compare 2 year differences from baseline among the 3 arms of the study; p < 0.001, ANOVA — 2 degree of freedom F-test from analysis of variance to compare 2 year differences from baseline among the 3 arms of the study, not adjusted for multiple comparisons among endpoints; 2 degree of freedom F-test from analysis of variance to compare 2 year differences from baseline among the 3 arms of the study; Mean Difference (Net) = 0.20, 95% CI 2-sided [-0.31 to 0.71]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare mean changes from baseline to year 2 among the 3 groups; Test type: Superiority; p = 0.002, ANOVA — This p-value is from a 2 degree freedom test of differences among the 3 groups; Mean Difference (Net) = 0.88, 95% CI 2-sided [0.37 to 1.39]

11. Secondary Outcome: Rigid Dietary Control
Description: Rigid control is characterized by an all-or-nothing inflexibility around dietary rules (e.g., strict calorie counting, with guilt following if calorie-dense foods are consumed) that is associated with poor weight outcomes and more binge eating (Westenhoefer, Stunkard, & Pudel, 1999). Scores range from 0 to 16 with higher scores reflecting greater rigid control.
  REF: Stunkard, A. J. M., S. (1988). Eating Inventory Manual. New York: Psychological Corporation.
Time Frame: Changes from baseline to 2 years
Measure: Mean (Standard Error); unit: 2 year changes in units on a scale
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 178 | 172 | 174
2 year changes in units on a scale | 0.35 (0.21) | 0.22 (0.21) | 1.75 (0.21)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; 2 degree F-test from analysis of variance applied to 2 year changes in scores from baseline; Test type: Superiority; p < 0.001, ANOVA — 2 degree of freedom F-test from analysis of variance; 2 degree of freedom F-test from analysis of variance to compare mean differences among arms; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.71 to 0.45]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare mean changes from baseline to 2 years among the 3 groups; Test type: Superiority; p < 0.001, ANOVA — This p-value is from the omnibus 2 degree of freedom test for mean differences among the 3 groups; Median Difference (Net) = 1.40, 95% CI 2-sided [0.82 to 1.98]

12. Secondary Outcome: General Health Index
Description: The General Health Index, a one-item question from the CDC's Health-Related Quality of Life measure (Measuring Healthy Days, 2000) required participants to report whether in general their health is excellent (1), very good (2), good (3), fair (4), or poor (5). Lower scores denotes better outcomes.
  Ref: Measuring Healthy Days. (2000). Atlanta, Georgia: Centers for Disease Control and Prevention
Time Frame: Changes from baseline to 2 years
Measure: Mean (Standard Error); unit: 2 year changes in units on a scale
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 178 | 172 | 174
2 year changes in units on a scale | 0.04 (0.06) | -0.04 (0.06) | -0.11 (0.06)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; 2 degree of freedom F-test from analysis of variance to compare 2 year differences in general health index values among the 3 arms; Test type: Superiority; p = 0.24, ANOVA — This p-value is from a 2 degree of freedom test for differences among the 3 arms; 2 degree of freedom test from analysis of variance to assess mean differences among the 3 arms; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.24 to 0.09]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare differences in changes from baseline to 2 years among the three arms; Test type: Superiority; p = 0.24, ANOVA — This p-value is from the 2 degree of freedom test of differences among the 3 arms; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.32 to 0.02]

13. Secondary Outcome: Mean Changes in High Density Lipoprotein Cholesterol (HDL-C)
Description: Mean changes in HDL-C from baseline to year 2 in (mg/dl) for compared among the 3 arms using analysis of variance
Time Frame: 2 years
Population: Mean changes among all participants with measurements at Year 2
Measure: Mean (Standard Error); unit: Mean Change from Baseline in mg/dl
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 158 | 154 | 159
Mean Change from Baseline in mg/dl | -0.09 (0.83) | 1.43 (0.82) | 2.12 (0.83)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Mean differences between baseline and year 2 were compared among the 3 arms using analysis of variance; Test type: Superiority; p = 0.16, ANOVA — This p-value is from a 2 degree of freedom F-test to compare the 3 arms using analysis of variance; Mean Difference (Net) = 1.52, 95% CI 2-sided [-0.77 to 3.81]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compared mean differences among the 3 groups; Test type: Superiority; p = 0.16, ANOVA — This p-value is from a 2 degree of freedom F test; Mean Difference (Net) = 2.21, 95% CI 2-sided [-0.09 to 4.51]

14. Secondary Outcome: Mean Changes in Low Density Lipoprotein Cholesterol (LDL-C)
Description: Mean changes between baseline and 2 years in low density lipoprotein cholesterol: LDL-c (mg/dl)
Time Frame: 2 years
Population: Mean changes from baseline among all participants with year 2 measures
Measure: Mean (Standard Error); unit: Mean change in LDL-C in mg/dl
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 158 | 154 | 159
Mean change in LDL-C in mg/dl | -0.01 (1.46) | 0.16 (1.44) | 1.43 (1.46)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Mean changes from baseline to year 2 among the 3 arms were compared using analysis of variance; Test type: Superiority; p = 0.75, ANOVA — This p-value is from a 2 degree of freedom F-test from analysis of variance; Mean Difference (Net) = 0.17, 95% CI 2-sided [-3.89 to 4.23]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare mean changes among the 3 groups; Test type: Superiority; p = 0.75, ANOVA — This p-value is from a 2 degree of freedom test; Mean Difference (Net) = 1.44, 95% CI 2-sided [-2.61 to 5.49] — No significant differences between groups 1 and 3

15. Secondary Outcome: Mean Change in Fasting Glucose From Baseline to 2 Years
Description: Mean change in fasting glucose from baseline to 2 years in mg/dl for all participants with year 2 measures
Time Frame: 2 years
Population: All participants with measurements at 2 years
Measure: Mean (Standard Error); unit: Mean change from baseline in mg/dl
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 158 | 154 | 159
Mean change from baseline in mg/dl | 1.48 (0.49) | 0.40 (0.49) | -0.18 (0.48)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Mean changes from baseline to year 2 among the 3 arms were compared using analysis of variance; Test type: Superiority; p = 0.05, ANOVA — This p-value is from a 2 degree of freedom F-test to compare the 3 arms within an analysis of variance; Mean Difference (Net) = -1.08, 95% CI 2-sided [-2.44 to 0.28] — No significant difference between groups 1 and 2
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare mean differences in changes from baseline to 2 years among the 3 groups; Test type: Superiority; p = 0.05, ANOVA — This p-value is from an F-test to compare differences among the 3 groups; Mean Difference (Net) = -1.66, 95% CI 2-sided [-3.00 to -0.32]

16. Secondary Outcome: Mean Change in Fasting Insulin From Baseline to 2 Years
Description: Mean change in fasting insulin (uU/ml) from baseline to 2 years
Time Frame: 2 years
Measure: Mean (Standard Error); unit: Mean changes at 2 years in uU/ml
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 158 | 154 | 159
Mean changes at 2 years in uU/ml | -0.27 (0.33) | -0.73 (0.33) | -1.48 (0.32)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Mean changes between baseline and year 2 were compared among the 3 arms using analysis of variance; Test type: Superiority; p = 0.03, ANOVA — This p-value is from a 2 degree of freedom F-test from an analysis of variance to assess differences among the 3 arms; Mean Difference (Net) = -0.46, 95% CI 2-sided [-1.37 to 0.45]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare mean differences from baseline to 2 years among the 3 groups; Test type: Superiority; p = 0.03, ANOVA — This p-value is from a 2 degree of freedom F-test to compare differences among the 3 groups; Mean Difference (Net) = -1.21, 95% CI 2-sided [-2.11 to -0.30]

17. Secondary Outcome: Depression Symptomatology
Description: Mean changes in the Center for Epidemiologic Studies Depression (CES-C) Scale. Reference: Turvey, C. L., Wallace, R. B., & Herzog, R. (1999). A revised CES-D measure of depressive symptoms and a DSM-based measure of major depressive episodes in the elderly. Int Psychogeriatr, 11(2), 139-148. 20 item questionnaire with a possible range of scores is zero to 60, and higher scores indicating the presence of more symptomatology.
Time Frame: 2 years
Population: All Participants with 2 year data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 178 | 172 | 174
units on a scale | 1.68 (0.50) | 0.60 (0.51) | 1.73 (0.51)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Mean differences from baseline to year 2 among the 3 arms were assessed using analysis of variance; Test type: Superiority; p = 0.20, ANOVA — This p-value is from a 2 degree of freedom F-test from an analysis of variance to assess mean differences among the 3 arms; Mean Difference (Net) = 1.08, 95% CI 2-sided [-0.84 to 3.00] — The 95% confidence interval for differences between groups 1 and 2 includes 0
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare differences among the 3 groups; Test type: Superiority; p = 0.20, ANOVA — This p-value is from an analysis of variance comparing all 3 groups; Mean Difference (Net) = -0.05, 95% CI 2-sided [-1.45 to 1.35] — The 95% confidence interval for differences between groups 1 and 3 includes 0

18. Secondary Outcome: Insulin Resistance
Description: We calculated homeostatic model assessment insulin resistance (HOMA-IR): fasting glucose in (mg/dl) * fasting insulin in (uU/mL).
Time Frame: Change from baseline to 2 years
Measure: Mean (Standard Error); unit: HOMA-IR
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 158 | 154 | 159
HOMA-IR | -0.03 (0.08) | -0.15 (0.08) | -0.33 (0.08)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; 2 degree of freedom F-test to compare mean 2 year differences among 3 arms; Test type: Superiority; p = 0.02, ANOVA — 2 degree of freedom F-test from analysis of variance, with no adjustment for multiple outcomes; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.34 to 0.10]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to compare mean differences in changes from baseline to 2 years among the 3 groups; Test type: Superiority; p = 0.02, ANOVA — This p-value is from a 2 degree of freedom test for differences among the 3 groups; Mean Difference (Net) = -0.30, 95% CI 2-sided [-0.52 to -0.08]

19. Secondary Outcome: Total Energy Dietary Intake Per Day (Kcals)
Description: Dietary intake was assessed using the 2005 Block Food Frequency Questionnaire (Block FFQ) at baseline and 2 years. This validated, quantitative 110-food item questionnaire is designed to assess relative intake of energy.
  REF: Block G, Woods M, Potosky A, Clifford C. Validation of a self-administered diet history questionnaire using multiple diet records. J Clin Epidemiol 1990; 43:1327-1335.
Time Frame: Changes from baseline to 2 years in kilocalories
Measure: Mean (Standard Error); unit: kilocalories
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 167 | 159 | 162
kilocalories | -134 (40) | -186 (41) | -185 (41)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; 2 degree of freedom F-test to compare mean differences among 3 arms in changes in kilocalories from baseline to year 2; Test type: Superiority; p = 0.58, ANOVA — 2 degree of freedom F-test to compare 3 arms with respect to 2-year changes in kilocalories; Mean Difference (Net) = -52, 95% CI 2-sided [-164 to 60]
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Analysis of variance was used to assess mean differences in 2 year changes in kilocalories intake among the 3 groups; Test type: Superiority; p = 0.58, ANOVA — This p-value is from a 2 degree of freedom F-test to compare differences among the 3 groups; Mean Difference (Net) = -50, 95% CI 2-sided [-162 to 61]

20. Secondary Outcome: Change in Waist Circumference (cm)
Description: Waist circumference will be measured using a Gulik tape measure and following a standardized protocol. Two measures of waist circumference will be taken; if the difference exceeds 1.0 cm, a third measure will be taken. Changes are measured from baseline to year 2.
Time Frame: Change from baseline to 2 years
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 159 | 154 | 159
centimeters | 0.21 (0.46) | -1.06 (0.47) | -2.21 (0.46)
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; 2 degree of freedom F-test from ANOVA to compare differences among 3 arms; Test type: Superiority; p = 0.001, ANOVA — 2 degree of freedom F-test from analysis of variance to compare changes in waist circumference from baseline among the three arms; No adjustment to degrees of freedom; Mean Difference (Net) = -1.27, 95% CI 2-sided [-2.55 to 0.02] — Difference between groups 1 and 2: 95% confidence interval includes 0
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Mean change in waist girth from baseline to year 2; Test type: Superiority; p = 0.001, ANOVA — The p-value is from a 2 degree of freedom F-test for differences among the 3 arms; Mean Difference (Net) = -2.42, 95% CI 2-sided [-3.69 to -1.14] — The 95% confidence interval for differences between groups 1 and 3 does not include 0

21. Secondary Outcome: Self-weighing
Description: Number of days per week the participant reports weighing themselves. This is divided into two groups: 1) more than once per week and 2) no more than once per week
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Small Behavior Changes | Large Behavior Changes
Number analyzed (Participants) | 152 | 145 | 153
Participants | 30 | 44 | 56
Statistical Analysis 1: Comparison: Control Group vs Small Behavior Changes; Logistic regression to compare differences among the 3 groups; Test type: Superiority — Chi-squared test to compare the percentage of participants reporting self-weighing more than once per week among the 3 arms; p = 0.004, Regression, Logistic — This is based on a 2 degree of freedom likelihood ratio test to compare differences among the 3 arms; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.04 to 3.02] — The 95% confidence interval for the odds ratio comparing the rates of self-weighing at year 2 between groups 1 and 2 excludes 0
Statistical Analysis 2: Comparison: Control Group vs Large Behavior Changes; Logistic regression analysis was used to compare the rates of daily self-weighing at 2 years among the 3 groups; Test type: Superiority; p = 0.004, Regression, Logistic — 2 degree of freedom likelihood ratio statistic to compare differences among the 3 arms; No adjustments; Odds Ratio (OR) = 2.35, 95% CI 2-sided [1.40 to 3.94] — The 95% confidence interval for the odds ratio comparing groups 1 and 3 excludes 0

22. Other Pre Specified Outcome: 6 Year Weight Changes
Description: Changes from baseline to year 6 in body weight
Time Frame: 6 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Event Data were collected on all participants from the time the participant signed the consent throughout the duration of the study (an average follow-up of 3 years). Participants were asked at each visit (scheduled to occur at months 4, 12, 24, 36, and 48 depending on when participants were enrolled relative to the end of follow-up) to report any medical events that occurred. Participants were also allowed to contact the clinic staff to report an adverse events at any intervening time
Description: Participants were asked about hospitalizations and any medical events at each study visit (4 months, 1 year, annually thereafter). Participants could also contact the study staff between visits to report an adverse event.
Arm/Group | Control Group | Self-regulation With Small Behavior Changes | Self-regulation With Large Behavior Changes
Serious Adverse Events (participants affected / at risk) | 4/202 | 11/200 | 9/197
Other Adverse Events (participants affected / at risk) | 119/202 | 118/200 | 109/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=202) | Self-regulation With Small Behavior Changes (N=200) | Self-regulation With Large Behavior Changes (N=197)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Gall bladder (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (2) — Stomach pain related to gallstones
Psychiatric (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (6) — One participant was hospitalized 3 times for depression. One participant was hospitalized twice for paranoid schizophrenia. One other participant was hospitalized once for depression.
Obstetric (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) | 0 (0)
Motor Vehicle Accident (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillectomy (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Tonsillectomy
E-coli bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Hospitalization for E-coli bacterial infection
Elective breast surgery (General disorders) | 1 (1) | 0 (0) | 0 (0) — Elective breast surgery
Stomach virus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Hospitalization for stomach virus
Benign mass (General disorders) | 0 (0) | 0 (0) | 1 (1) — Outpatient surgery for benign mass on left maxillary sinus
Syncope (General disorders) | 0 (0) | 0 (0) | 1 (1) — Syncope led to fall and hospitalization for concussion
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Hospitalization for Crohn's disease
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Rheumatoid arthritis - increased pain following pregnancy -- condition was present 10 years prior to study entry
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=202) | Self-regulation With Small Behavior Changes (N=200) | Self-regulation With Large Behavior Changes (N=197)
Cardiovascular (Cardiac disorders) | 3 (3) | 7 (7) | 7 (7)
Muscoskeletal (Musculoskeletal and connective tissue disorders) | 55 (65) | 50 (63) | 45 (51)
Diabetes (Endocrine disorders) | 2 (3) | 1 (1) | 0 (0)
Gall bladder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Psychiatric (Psychiatric disorders) | 16 (17) | 18 (20) | 16 (18)
Ashthma Attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Obstetric (Pregnancy, puerperium and perinatal conditions) | 15 (21) | 13 (15) | 10 (13)
Weight loss related (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Motor vehicle accident (General disorders) | 26 (30) | 28 (31) | 27 (30)
Other (General disorders) | 56 (68) | 40 (48) | 54 (64)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No